CLINICAL TRIAL: NCT02235753
Title: High-Intensity Exercise Training in Cardiac Rehabilitation After Acute Coronary Event - Randomized Controlled Trial
Brief Title: High-intensity Exercise After Acute Cardiac Event (HITCARE)
Acronym: HITCARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was stopped due to lack of funding.
Sponsor: Kuopio Research Institute of Exercise Medicine (Other)
Collaborators: Social Insurance Institution, Finland (Other); Kuopio University Hospital (Other); University of Eastern Finland (Other); University of Basel (Other)
Responsible Party: Principal Investigator, Rainer Rauramaa, Professor, Kuopio Research Institute of Exercise Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1072011
Record Dates: First submitted 2014-09-03; First posted 2014-09-10 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2015-12

CONDITIONS: Unstable Angina Pectoris; Acute Myocardial Infarction; Recurrent Myocardial Infarction
MeSH Terms: conditions — Angina, Unstable; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High-intensity interval training, HIT-S (Experimental): High-intensity aerobic interval training, short interval (HIT-S)
  Interventions: Behavioral: High-intensity aerobic interval training, short interval
- High-intensity interval training, HIT-L (Experimental): High-intensity aerobic interval training, long interval (HIT-L)
  Interventions: Behavioral: High-intensity aerobic interval training, long interval
- Usual care (No Intervention): control group

INTERVENTIONS:
Behavioral: High-intensity aerobic interval training, short interval — The intensity of HIT-S sessions (cycle ergometer) will be increased during 3 to 6 months from 60% of VO2peak to 100% which will be the target intensity from 6 to 12 months. The protocol includes four 6 min sets consisting of 15 sec exercise followed by 15 sec passive recovery separated with 3 min passive recovery between sets. Exercise session will last ca. 40 min, with 12 min of HIT, warm-up and recovery. The intensity of the 15 seconds exercise bouts will be based on VO2peak at baseline and after 6 months. Meanwhile, the estimated VO2peak from the submaximal test will be used to adjust the training intensity in HIT sessions. Training will be conducted in a group of 1-3 HIT-S patients with ECG monitoring and supervised by physician.
  Arms: High-intensity interval training, HIT-S
Behavioral: High-intensity aerobic interval training, long interval — The intensity of HIT-L sessions (cycle ergometer) will be increased during 3 to 6 months from 60% of VO2peak to 90% which will be the target intensity from 6 to 12 months. The protocol includes four 3 min exercise bouts with a 4 min recovery (pedaling at 0 W) between bouts. Exercise session will last ca. 40 min, with 12 min of HIT, warm-up and recovery. The intensity of the 3 min exercise bouts will be based on VO2peak at baseline and after 6 months. Meanwhile, the estimated VO2peak from the submaximal test will be used to adjust the training intensity in HIT sessions. Training will be conducted in a group of 1-3 HIT-L patients with ECG monitoring and supervised by physician.
  Arms: High-intensity interval training, HIT-L

SUMMARY:
Despite the well-known health benefits of physical exercise in the prevention of chronic diseases, less attention has been focused on the use of physical exercise as an essential part of good treatment for chronic disease. The aims of the study are to investigate the feasibility, medical effects, cost-effectiveness, and social perspectives of the individualized exercise-based rehabilitation [2 different high-intensity training (HIT) protocols combined with usual care (UC)] after acute coronary artery disease (CAD) event. The medical aim is to study mediating mechanisms of the physiological, biochemical and molecular effects of exercise training on the clinical outcomes. The aim of the health-economic evaluation is to assess the changes in the Health-Related Quality of Life (HRQL) and health care related costs for estimating the cost-effectiveness of HIT-based exercise rehabilitation. The purpose of the sociological analysis is to find out the social processes which make possible the emergence of the desired welfare effects.

DETAILED DESCRIPTION:
The study population consists of patients living in the city of Kuopio or Siilinjarvi area in Eastern Finland, who have been treated in Kuopio University Hospital because of acute CAD event. After baseline measurements, the patients will be randomized into one of the 3 groups: short interval HIT protocol (HIT-S), long interval HIT protocol (HIT-L) or UC group. The intervention will be 12 months per patient and the expected duration of the whole study (intervention data collection) is estimated to be 4 years. In addition, all groups will have annual follow-up examinations scheduled up to 60 months after initiation of the intervention phase. The patients recruited for the study will be 750, a total of 250 patients per study group.

All measurements related to intervention will be performed at Kuopio Research Institute of Exercise Medicine. Examinations concerning myocardial structure and perfusion will be done at Turku PET Center (subsample).

The study complies with the Helsinki declaration, follows good clinical practice. Patient safety will follow normal medical practice. The intervention is not anticipated to cause health risks apart from the conventional treatment. All participants will be provided with diverse individualized information about their health and physical performance. The research methods employed in the study are safe. Physician and nurse will be present at each occasion when physically strenuous measurements are performed and careful provisions for appropriate first aid will be made. The measurements assessing cardiorespiratory and muscular fitness will involve hard effort and it is not unusual to feel innocent muscle pain for a few days after measurements demanding maximal effort. The other potential acute complications may include accidents (e.g. injuries due to slipping or falling) and medical emergencies like acute myocardial infarction.

Study hypotheses:

1. Short (15 sec) and long interval (3 min) high-intensity aerobic interval training (HIT) combined with resistance training after acute CAD event are equally effective in improving cardiorespiratory fitness compared with UC.
2. Despite higher unit costs, the differences in health-related quality of life effects are so large that both HIT interventions are cost-effective compared with UC.
3. Patient's experiences and interpretation of HIT exercise as well as different social processes during rehabilitation explain the cost-effectiveness of the rehabilitation.
4. Patient groups who will or will not benefit of HIT interventions can be identified and predicted.

ELIGIBILITY:
Inclusion Criteria:

* hospital care after acute CAD event (ICD-10 codes I20.0-I22)
* age 40-80 years
* signed informed consent form

Exclusion Criteria:

* conditions preventing regular exercise training
* severe/malignant disease (life expectancy <12 months)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-12; Primary Completion 2016-11-14 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness as assessed by peak oxygen uptake (VO2peak) | Baseline, 6 and 12 months

SECONDARY OUTCOMES:
Incremental health care cost/quality-adjusted life-year-relation | Baseline, 6 and 12 months
Social processes explaining adherence and motivation to exercise rehabilitation | Baseline, 6 and 12 months
  Social analysis will be performed by specific questionnaires and interviews. Subjective perceptions on the social mechanisms impacting on health and well-being as a part of the rehabilitation processes will be also be modelled using comparative causal mapping techniques (CMT) (See http://www.uef.fi/fi/cmap3).
Total costs of the use of health care services | Baseline, 6 and 12 months
  The use of total health services will be assessed by diary, questionnaire and from registers (national, hospital district and domicile health center).
Utilization of health care resources | Baseline, 6 and 12 months
Change in health-related quality of life | Baseline, 6 and 12 months

OTHER OUTCOMES:
Change in ergospirometer variables | Baseline, 6 and 12 months
Change in muscular performance | Baseline, 6 and 12 months
Change in daily energy expenditure | Baseline, 6 and 12 months
Sleeping time | Baseline, 6 and 12 months
Sitting time | Baseline, 6 and 12 months
Dietary habits | Baseline, 6 and 12 months
  Measured by food frequency questionnaire
Change in chest pain symptoms, exercise induced angina or ischemia | Baseline, 6 and 12 months
  Composite measure based on anamnesis and ECG
Change in antianginal and other medication | Baseline, 6 and 12 months
Hospitalization due to cardiovascular causes | Baseline, 6 and 12 months
Change in vascular risk factors | Baseline, 6 and 12 months
Progression of peripheral atherosclerosis | Baseline, 6 and 12 months
Change in cognitive function | Baseline and 12 months
Change in depressive symptoms | Baseline, 6 and 12 months
Intervention related adverse events | Throughout the intervention phase
Change in myocardial blood flow capacity and left ventricular function | Baseline and 12 months
Change in myocardial blood flow at rest and during adenosine infusion | Baseline and 12 months
Change in myocardial blood flow reserve | Baseline and 12 months
Change in left ventricular ejection fraction | Baseline and 12 months
Change in left ventricular longitudinal peak systolic strain | Baseline and 12 months
Change in left mitral annular diastolic tissue velocity | Baseline and 12 months
Change in autonomic nervous system control of cardiac function | Baseline and 12 months
Change in body composition | Baseline, 6 and 12 months
  Measured by bioimpedance
Change in anthropometric measures | Baseline, 6 and 12 months
  Measured by body weight, body height, waist circumference, and hip circumference.
  Body mass index and waist to hip ratio will be calculated.
All-cause death | Baseline, 6 and 12 months; annual follow-up up to 60 months
Cardiovascular death | Baseline, 6 and 12 months; annual follow-up up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Rauramaa, professor, Principal Investigator — Kuopio Research Institute of Exercise Medicine
Locations (1):
- Kuopio Research Institute of Exercise Medicine, Kuopio, Finland